CLINICAL TRIAL: NCT06152406
Title: Safety and Efficacy of Distal His Bundle Pacing Compared to Right Ventricular Pacing in Patients With Symptomatic Atrial Fibrillation Undergoing AV Node Ablation With Evidence of Heart Failure, a Randomised Control Study
Brief Title: Ablate and Pace HIS Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 153856
Record Dates: First submitted 2023-09-21; First posted 2023-11-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: HIS Bundle Pacing; Atrial Fibrillation
Keywords: HIS Bundle Pacing; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right Ventricular Only Pacing (Active Comparator): All study participants will have an RV lead inserted, but this arm will have an RV lead only.
  Interventions: Procedure: Ablation and Pacemaker Implantation
- HIS Bundle Pacing (Other): Participants in this group will have HIS bundle pacing, but in addition will have an RV lead inserted that will serve as a backup alternative in the event HIS bundle pacing is not effective.
  Interventions: Procedure: Ablation and Pacemaker Implantation

INTERVENTIONS:
Procedure: Ablation and Pacemaker Implantation — All patients will be implanted with a pacemaker device with one lead positioned in right ventricle (control arm only) and an additional lead will be positioned on the distal (ventricular) HIS bundle if in intervention arm. All patients will undergo ablation.

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia, and estimates suggest its prevalence is increasing. Despite the advances in AF ablation strategies, the outcome of ablation procedures in persistent AF is still unsatisfactory. In addition, many patients are not candidates for ablation due to advanced age, comorbidities and previous failed ablation procedures.

It is well known that there is no mortality benefit from rhythm versus rate control strategy in AF, therefore the increased number of AV node ablation and pacemaker insertion for patients with symptomatic AF with uncontrolled heart rate. Following AV node ablation, it is understandable that these patients will be paced 100% of the time where the value of physiological pacing will be at its most.

The current standard practice is to pace the right ventricle for this cohort of patients unless they have severe LV systolic dysfunction when a biventricular pacing might be recommended. Previous data showed that RV pacing only can lead to deterioration of LV function, worsening of heart failure symptoms and increased mortality.

HIS bundle pacing is a novel technique of pacing through placing the pacemaker lead on the junction box between the top and bottom chamber of the heart. This will allow the utilisation of the normal/intrinsic HIS Purkinjie (eclectic cables) to stimulate the ventricles. This can offer a physiological pacing modality and reduce pacing induced cardiomyopathy specially in pacing dependent pacing.

The Ablate and Pace HIS Study proposes that the new method of HIS pacing is safe, effective and superior to the existing method of RV pacing in patients with atrial fibrillation who demonstrate signs of heart failure.

DETAILED DESCRIPTION:
The Ablate and Pace HIS Study is a single-centre, prospective randomised single-blinded study, recruiting a sub-population of patients with AF who are deemed not fit for rhythm control strategy. These patients have been referred for a pacemaker implant and AVN node ablation as a symptomatic rate control option.

The study aims to randomise a total of 100 participants into either the RV only pacing arm or the HBP arm. All patients will be implanted with a pacemaker device with one lead positioned in the right ventricle, and only in the HBP arm will an additional lead be positioned on the distal HIS bundle in order to obtain direct HIS-bundle capture. The RV lead will be only be used as a back-up option for the HBP arm if needed.

Participants will undergo AVN ablation either at the same setting or 4-6 weeks later according to clinical indication and operator preference. A double-blinded design will then be employed to investigate the effect of HIS pacing. Endpoint measurements will be taken at Baseline, 4 weeks, 6 months and 12 months post randomisation. Treatment allocation will be blinded to the patients and endpoint assessor. All participants will be informed of their allocated treatment arm at the end of their 12 month follow up visit.

Funding has been provided by Medtronic. The study Sponsor is University Hospitals of Leicester.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Symptomatic AF, New York Heart Association (NYHA) class II-IV
* Willing to consent for the study
* AF regardless type, deemed not suitable for rhythm control strategy that has been referred for AVN ablation with one of the following:

  1. Impaired LV function, EF <50 %. And or
  2. Raised N-Terminal Pro B-type Natriuretic Peptide ( NT-ProBNP) >365 ng/L

Exclusion Criteria:

* Patient who has already got a pacemaker in situ
* Known severe LVSD when biventricular device is the thought to be the preferred pacing modality
* Females in child bearing period
* Lack of capacity to consent
* Other serious medical condition with life expectancy of less than 1 year
* Less than 18 years
* Unwilling to consent for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with 20% improvement in 6 minutes-walk distance, AFEQT questionnaire score, and number of steps and distance walked per day assessed by a Fitbit smart watch | 12 months
  20% improvement in all 3 areas

SECONDARY OUTCOMES:
Improvement of LV function, LVESV assessed by echocardiogram | 12 months
  Improvement of LV function, LVESV assessed by echocardiogram
Change in NT-ProBNP level | 12 months
  Change in NT-ProBNP level
Incidence of hospitalisation for heart failure, need for device upgrade to biventricular pacemaker or mortality | 12 months
  Incidence of hospitalisation for heart failure, need for device upgrade to biventricular pacemaker or mortality
Pacing parameters | 12 months
  RV threshold/HIS bundle lead will be checked, and this will be documented if it has changed.
Fluoroscopy time during the device insertion | During device insertion
  Fluoroscopy time during the device insertion
Safety consideration: rate of infection, lead failure, displacement or the need for a repeat procedure | 12 months
  Safety consideration: rate of infection, lead failure, displacement or the need for a repeat procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided